CLINICAL TRIAL: NCT05167214
Title: The Acute Effect Of Different Kinesiological Tape Application On Pain, Functional Performance And Trunk Endurance In Young Adults With Chronic Back Pain
Brief Title: The Acute Effect Of Different Kinesiological Tape
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Collaborators: Okan University (Other)
Responsible Party: Principal Investigator, mustafa gulsen, assocc.prof., Baskent University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: BaskentUU
Record Dates: First submitted 2021-10-19; First posted 2021-12-22 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: Chronic Back Pain
Keywords: Kinesiology Taping; Visual Pain Scale; Oswestry; Chronic Low Back Pain; Functional Performance

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Star tape (Experimental): Group 1 ( n=35) was applied with the star technique. Visual Analogue Scale (VAS) to evaluate pain before taping, immediately after taping and 4 days after taping, Oswestry low back pain disability scale (OLBPDS) to assess disability level, Lumbar Flexion Repeat Speed Test, Sit-and-Stand Test to evaluate functional performance in both groups. Biering Sorenson Test was applied to evaluate the forward bending test with weight and trunk endurance. Individuals in both groups were told to continue with their daily lives while on the tapes. It was stated that the bands should stay on the applied area for 4 days, that they can have a bath while the bands are on, and that if the bands are uncomfortable or excessive itching on the skin, the individuals can remove the bandage with an oily solution. No itching, redness, or allergic reactions was observed in either group.
  Interventions: Device: The Acute Effect Of Different Kinesiological Tape Application On Pain, Functional Performance And Trunk Endurance In Young Adults With Chronic Back Pain
- I Tape (Placebo Comparator): Group 2 (n=35) was applied in the form of I tape. Visual Analogue Scale (VAS) to evaluate pain before taping, immediately after taping and 4 days after taping, Oswestry low back pain disability scale (OLBPDS) to assess disability level, Lumbar Flexion Repeat Speed Test, Sit-and-Stand Test to evaluate functional performance in both groups. Biering Sorenson Test was applied to evaluate the forward bending test with weight and trunk endurance. Individuals in both groups were told to continue with their daily lives while on the tapes. It was stated that the bands should stay on the applied area for 4 days, that they can have a bath while the bands are on, and that if the bands are uncomfortable or excessive itching on the skin, the individuals can remove the bandage with an oily solution. No itching, redness, or allergic reactions was observed in either group.
  Interventions: Device: The Acute Effect Of Different Kinesiological Tape Application On Pain, Functional Performance And Trunk Endurance In Young Adults With Chronic Back Pain

INTERVENTIONS:
Device: The Acute Effect Of Different Kinesiological Tape Application On Pain, Functional Performance And Trunk Endurance In Young Adults With Chronic Back Pain — The Acute Effect Of Different Kinesiological Tape Application On Pain, Functional Performance And Trunk Endurance In Young Adults With Chronic Back Pain

SUMMARY:
This study aims to compare the acute effects of different kinesiology tapes on pain, functional performance and trunk endurance in young adults with chronic low back pain. Seventy young adults with chronic low back pain between the ages of 18-40 were included in our study. The individuals included in our study were divided into two groups by a simple randomization method. Star-shaped kinesiology taping was applied to the 1st group, and I-shaped kinesiology taping was applied to the 2nd group. The demographic and physical characteristics of the individuals who agreed to participate in the study were recorded. Visual Analogue Scale (VAS) to evaluate pain before taping, immediately after taping and 4 days after taping, Oswestry low back pain disability scale (OLBPDS) to assess disability level, Lumbar Flexion Repeat Speed Test, Sit-and-Stand Test to evaluate functional performance in both groups. Biering Sorenson Test was applied to evaluate the forward bending test with weight and trunk endurance.

DETAILED DESCRIPTION:
Star-shaped kinesiology taping was applied to the 1st group, and I-shaped kinesiology taping was applied to the 2nd group. The demographic and physical characteristics of the individuals who agreed to participate in the study were recorded. Visual Analogue Scale (VAS) to evaluate pain before taping, immediately after taping and 4 days after taping, Oswestry low back pain disability scale (OLBPDS) to assess disability level, Lumbar Flexion Repeat Speed Test, Sit-and-Stand Test to evaluate functional performance in both groups. Biering Sorenson Test was applied to evaluate the forward bending test with weight and trunk endurance.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 18-40 who accept participating in the research,
* low back pain for at least 3 months,
* have no perception problems
* can cope well,
* individuals who regularly come to the controls and evaluations of the physical therapy program.

Exclusion Criteria:

* undergone spinal surgery,
* have complain of low back pain due to inflammatory, tumoral, metabolic cause, orthopedic (pes planus, genu varum, genu valgum, scoliosis, etc.) or neurological (Multiple Sclerosis, Stroke, etc.) problems that prevent treatment, spine or lower back pain.
* have extremity surgery,
* have another musculoskeletal disorder affecting the lower extremity,
* pregnancy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2021-03-25 (Actual); Study Completion 2021-05-10 (Actual)

PRIMARY OUTCOMES:
Kinesiological Tape Application | 4 days
  The individuals included in our study were divided into two groups by a simple randomization method. Star-shaped kinesiology taping was applied to the 1st group, and I-shaped kinesiology taping was applied to the 2nd group.

SECONDARY OUTCOMES:
Visual Analogue Scale | 4 days
  Patients were asked to mark the pain they felt on a 10 cm scale between '0' (I have no pain) and '10' (I have unbearable pain), the distance between the marked point and the starting point was measured and recorded as data.
Oswestry Scale | 4 days
  The Turkish version of the Oswestry Scale was applied to individuals to measure the low back pain disability level of the individuals. The study on the validity of the questionnaire was conducted by Yakut et al. In this scale, there are 10 questions evaluating various activities of daily living and 6 options for each question with a score between 0 and 5. 0-4 points as no disability, 5-14 points as mild, 15-24 points as moderate, 25-34 points as severe and 35-50 points as complete functional disability. The lowest score obtained from the scale is 0, and the highest score is 50. A score of 50 indicates the maximum level of functional disability.
Lumbar Flexion Repeat Speed Test | 4 days
  To evaluate functional performance. Before starting the test, warm-up flexion was performed 3 times, and the individual was asked to bend forward 10 times as fast as he could, while standing and both heels together, and to straighten as fast as he could again. The chronometer was started with the start command, the chronometer was stopped after 10 consecutive flexion and extension were completed, and the elapsed time was recorded in seconds.
Sit-and-Stand Test | 4 days
  To evaluate functional performance is the Sit-Up test (OKHT). After sitting on a chair, the individual was asked to get up and sit down as fast as he could 5 times, the chronometer was started with the start command, and the elapsed time was recorded in seconds after the last sitting was completed.
Biering Sorenson Test | 4 days
  to assess the trunk endurance. Trunk Extensor Muscle Endurance (Biering-Sorensen Test): The individual was prone placed by hanging from the bed from the anterior superior of the spina iliaca, and was fixed at the gastrocnemius muscle level. He was asked to keep his torso parallel to the ground by clasping his hands on the chest. The time that parallelism was maintained was recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Okan University, Istanbul, Turkey (Türkiye)